CLINICAL TRIAL: NCT05103917
Title: An Open Label, Phase Ib/II Trial to Study the Safety, Tolerability and Antitumor Activity of X4P-001 in Combination With Toripalimab in Patients With Locally Advanced or Metastatic Triple Negative Breast Cancer (TNBC)
Brief Title: A Study to Assess the Safety, Tolerability and Antitumor Activity of X4P-001 in Combination With TNBC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X4P-001-201
Record Dates: First submitted 2021-09-25; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — mavorixafor; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- X4P-001-201 (Experimental): trial to Study the Safety, Tolerability and Antitumor Activity of X4P-001 in Combination with Toripalimab in Patients with Locally Advanced or Metastatic Triple Negative Breast Cancer (TNBC)
  Interventions: Drug: X4P-001

INTERVENTIONS:
Drug: X4P-001 — CXCR4 inhibitor
  Other Names: Toripalimab Injection

SUMMARY:
Objectives Phase 1b

Primary Objectives:

To evaluate the safety and tolerability of X4P-001 combined with toriplimab in patients with locally advanced or metastatic TNBC

Secondary Objectives:

1. To characterize the pharmacokinetics (PK) profile of X4P-001 alone or combined with toriplimab
2. To characterize the antitumor activity of X4P-001 in combination with toriplimab in patients with locally advanced or metastatic TNBC(according to RECIST 1.1)
3. To characterize the overall survival of X4P-001 in combination with toriplimab in patients with locally advanced or metastatic TNBC
4. To characterize the immunogenicity of toriplimab when administrated in combination with X4P-001

DETAILED DESCRIPTION:
Exploratory Objectives:

1. To explore selected biomarkers in peripheral blood and tumor samples that potentially correlate with clinical response to X4P-001 and toriplimab combination treatment
2. To characterize the antitumor activity of X4P-001 in combination with toriplimab in patients with locally advanced or metastatic TNBC(according to iRECIST 1.1)

ELIGIBILITY:
Inclusion Criteria:

* 1. Female, age 18 ~ 75 (including both ends, or other age range required by local regulations or IRB).

  2. Patients must have histological confirmed locally advanced or metastatic TNBC:

  a) The primary or metastatic lesions were pathologically confirmed to be triple negative, that is, negative for ER, PR and HER-2. Negative ER and PR are defined as ER < 1% positive and PR < 1% positive. HER-2 negative is defined as: immunohistochemical detection of HER-2 (-) or (1 +), HER-2 (2 +) must be tested for FISH and the result is negative, HER-2 (1 +) can be selected for FISH test and the result is negative, and metastatic pathology is preferred b) Patient must have at least 1 measurable lesion (by RECIST V1.1) c) Patient must progress after first-line and not more than second-line systematic treatment d) Patient must agree to undergo a tumor biopsy in the study e) Previous tumor tissue samples that meet the requirements should be provided during the screening period, or tumor biopsies should be performed before the first treatment.

  3. ECOG performance status 0~1 4. Life expectancy ≥ 12 weeks 5. Adequate organ function and bone marrow function as indicated by the following screening assessments performed within 14 days before the first dose of study drug (without blood transfusion or medication with stimulation factors within 14 days before 1st dose) :
  1. Absolute neutrophil count (ANC) ≥1.5×109/L
  2. Platelet count (PLT) ≥100×109/L
  3. Hemoglobin (Hb) ≥90 g/L
  4. Total bilirubin (TBIL) ≤1.5×ULN
  5. Aspartate transaminase (AST) and alanine transaminase (ALT), ≤2.5 ×ULN (for the patient with liver metastasis in escalation part or patient in expansion part: AST and AST ≤5×ULN)
  6. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (Crcl) ≥50mL/min based on Cockcroft-Gault formula 6. Female patients of childbearing potential must agree to use effective methods of birth control during the study and for up to 6 months after the last dose of study drug. Non-surgically sterilized female patients of childbearing potential must be in non-lactation period, and have a negative β-HCG test result within 7 days before first administration.

     7. Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.

     Exclusion Criteria:
* 1. Patients who are known to be allergic to any component of X4P-001 or triplizumab or have previously developed severe allergic reactions, rapid allergic reactions or other hypersensitivity to peptides, chimeric or humanized antibodies, fusion proteins 2. Patients who suffer from other malignant tumors within 5 years before enrollment (except: radical cervical carcinoma in situ or non-melanoma skin cancer; second primary cancer that has been cured and has no recurrence within five years; the researchers believe that both primary cancers can benefit from this study; the researchers have clearly confirmed which primary tumor source the metastatic focus belongs to).

  3. Patients with primary central nervous system malignant tumor; patients with central nervous system metastasis who failed local treatment; (patients with asymptomatic brain metastasis, or patients with stable clinical symptoms and without steroids and other treatment for brain metastasis for more than 28 days can be included in the group. ).

  4. Patients who use cytochrome P450 (CYP) 3A4, strong 2D6 inhibitors or inducers (see 12.4, including prohibited foods) and antacids before the first use, and the last use is less than 14 days or 5 half-lives from the first use, whichever is the shorter.

  5. Patient who RANKL ligand inhibitors were used within 1 month before the first administration of the study drug or are expected to be used during the study period (e.g. deschumab, etc.) 6. Patients who systemic immunosuppressive drugs (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, etc.) are used within 2 weeks prior to the first administration of research drugs, or systemic immunosuppressive drugs are known to be required in the course of research treatment, unless:
  1. Patients who receive short-term, low-dose systemic immunosuppressive drugs or patients who receive one-time systemic immunosuppressive drug pulse therapy (such as corticosteroids for 48 hours for the treatment of contrast medium allergic reactions, single use of cyclophosphamide during induction of tumor therapeutic vaccine)
  2. Patients who receive corticosteroids in the treatment of chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids in the treatment of orthostatic hypotension or adrenal insufficiency are allowed to enter the group 7. Previous anti-cancer therapy prior to initiation of study treatment: major surgery (except palliative therapy), radiotherapy (bone-marrow exposure >30%);routine chemotherapy, targeted therapy, immunotherapy is less than 4 weeks (chemotherapy with nitrosourea or mitomycin <6 weeks); endocrine therapy within ≤ 5 half-life or ≤ 14 days (whichever is shorter).

     8. Patients who are unable to take oral drugs or there are factors that significantly affect oral drug absorption, such as gastric remnant dysfunction after previous total gastrectomy or subtotal gastrectomy, short bowel syndrome after small bowel resection, active diarrhea or irritable bowel syndrome requiring drug treatment, etc.

     9. Patients with previous organ transplants 10. Patients with definite active infection or fever of unknown origin > 38.3 ℃ within 4 weeks before receiving the first study drug and were treated with oral or intravenous antibiotics.

     11. Patients who had previously participated in other clinical studies were included in the original clinical study and less than 28 days after the first administration of the drug in this study.

     12. Patients whose adverse events caused by previous antineoplastic therapy did not recover to ≤ grade 1 (CTCAE5.0) (except for alopecia, vitiligo, ≤ grade 2 neurotoxicity and other events that researchers believe do not affect the safety evaluation of patients and research drugs).

     13. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

  a) New York Heart Association class III or IV congestive heart failure, unstable angina, or myocardial infarction within 6 months before administration of the study drug; b) Clinically significant cardiac arrhythmia requiring active therapy; c) Uncontrolled hypertension; d) Left ventricle ejection fraction<50%; e) Prolongation of QTcF (average of three times of examine, male > 450 ms, female > 470 ms) (Note: QTc interval corrected by Frederica's formula) at screening, and other ECG abnormalities with clinical significant by the judge of the investigator.

  14. Patients with a history of interstitial pneumonia 15. Patients were positive for (HIV) antibody of human immunodeficiency virus, (HCV) antibody of hepatitis C virus and (TP) antibody of Treponema pallidum, and (HBV) surface antigen of hepatitis B virus was positive and HBVDNA ≥ 1000IU/ml. The subjects are in active stage of tuberculosis; (antiviral therapy is allowed during the trial of subjects with positive (HBV) surface antigen of hepatitis B virus).

  16. Any other clinically significant comorbidities, such as respiratory, metabolic, congenital, endocrine or central nervous system disease, or any other medical conditions, mental disturbances or social determinants, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-11-24 (Estimated); Study Completion 2023-05-21 (Estimated)

PRIMARY OUTCOMES:
CT | Screening
  resist 1.1 evaluation
CT | C3D1 (12 weeks)
  resist 1.1 evaluation

CONTACTS AND LOCATIONS:
Overall Officials: J L Zheng, Director, Study Director — Abbisko Therapeutics Co, Ltd
Locations (1):
- Shang hai Tumor Hospital, Shanghai, Shanghai Municipality, China